CLINICAL TRIAL: NCT02681081
Title: Optimizing Chronic Pain Treatment With Enhanced Neuroplastic Responsiveness
Acronym: OPTIMIZE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Pain Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB201400913; OCR15965 (Other: University of Florida)
Record Dates: First submitted 2016-02-02; First posted 2016-02-12 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Pain; Osteoarthritis
Keywords: Neuroplasticity
MeSH Terms: conditions — Pain; Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Other): For sessions 2 through 4, maintain normal eating patterns.
  Interventions: Other: Control
- Glucose Administration (Active Comparator): For sessions 2 through 4, participants will fast for two hours prior to each session and consume 25-30 g of glucose at the start of each session.
  Interventions: Other: Glucose Administration
- Intermittent Fasting (Active Comparator): For sessions 2 through 4, participants will fast for 16 hours prior to the session (no food or beverages other than non-caloric beverages or coffee after 6 or 7 pm the evening prior).
  Interventions: Other: Intermittent Fasting

INTERVENTIONS:
Other: Glucose Administration — For sessions 2 through 4, participants will fast for two hours prior to each session and consume 25-30 g of glucose at the start of each session.
  Arms: Glucose Administration
Other: Intermittent Fasting — For sessions 2 through 4, participants will fast for 16 hours prior to the session (no food or beverages other than non-caloric beverages or coffee after 6 or 7 pm the evening prior).
  Arms: Intermittent Fasting
Other: Control — Normal food intake
  Arms: Control

SUMMARY:
The purpose of the study is to identify non-invasive strategies that will optimize the neurobiological environment and improve learning and memory in the treatment of chronic pain. The overall aims of the current proposal are to determine if food restriction and/or glucose administration in conjunction with a relaxation/guided imagery exercise will result in neurophysiological changes and functional improvements compared to the relaxation/guided imagery exercise alone.

DETAILED DESCRIPTION:
Up to sixty adults with chronic knee pain with or/at risk of knee osteoarthritis will be randomized to one of three groups: food restriction (20 participants), glucose administration (20 participants), or control (20 participants). Participants will attend four sessions over a two to three week period.

ELIGIBILITY:
Inclusion Criteria:

* Adults with chronic knee pain with or/at risk of knee osteoarthritis

Exclusion Criteria:

* Concurrent medical condition that could confound outcome measures or limit the ability to participate completely in the protocol including: neurological conditions (Parkinson's disease, multiple sclerosis, and/or seizures)
* History of a head injury or stroke
* Diabetes or taking medications to control blood sugar
* Mental health issues resulting in hospitalization or outpatient treatment in the past year, and/or psychotropic medication use
* Current issue or history of treatment for alcohol or other substance abuse
* Cognitive function < or = 22 on the Mini-Mental Status Exam
* Pregnancy
* A baseline fasting blood sugar (plasma glucose > 7mmol/L) or persisting blood pressure >150/95.
* Heart condition such as a prior heart attack, heart surgery (including a stent), frequent chest pain or heart failure
* Inability to complete the EEG portion of the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Change in Neurophysiological measures | baseline and 3 weeks
  Electroencephalogram (EEG) amplitude measures.

SECONDARY OUTCOMES:
Change in Clinical Pain measure - Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline and 3 weeks
  Measure of lower extremity pain and function in persons with knee OA.
Change in Experimental Pain measure - Temporal summation of punctate mechanical stimuli | baseline and 3 weeks
  Quantitative sensory testing measure.
Change in Level of Distress measure - Perceived Stress Scale | baseline and 3 weeks
  Measure of perceived stress.
Change in Affect Measure - Positive and Negative Affect Schedule (PANAS) | baseline and 3 weeks
  Measure of positive and negative affect.

OTHER OUTCOMES:
Change in Recall and Recognition measures - Hopkins Verbal Learning Test (HVLT) | baseline and 3 weeks
  Measure of verbal learning/memory

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly T Sibille, PhD, Principal Investigator — University of Florida
Locations (1):
- Institute of Aging, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith MA, Riby LM, Eekelen JA, Foster JK. Glucose enhancement of human memory: a comprehensive research review of the glucose memory facilitation effect. Neurosci Biobehav Rev. 2011 Jan;35(3):770-83. doi: 10.1016/j.neubiorev.2010.09.008. Epub 2010 Sep 29. PMID 20883717
- [Background] Hensch TK, Bilimoria PM. Re-opening Windows: Manipulating Critical Periods for Brain Development. Cerebrum. 2012 Jul;2012:11. Epub 2012 Aug 29. PMID 23447797
- [Background] Martin B, Mattson MP, Maudsley S. Caloric restriction and intermittent fasting: two potential diets for successful brain aging. Ageing Res Rev. 2006 Aug;5(3):332-53. doi: 10.1016/j.arr.2006.04.002. Epub 2006 Aug 8. PMID 16899414
- [Background] Cramer SC, Sur M, Dobkin BH, O'Brien C, Sanger TD, Trojanowski JQ, Rumsey JM, Hicks R, Cameron J, Chen D, Chen WG, Cohen LG, deCharms C, Duffy CJ, Eden GF, Fetz EE, Filart R, Freund M, Grant SJ, Haber S, Kalivas PW, Kolb B, Kramer AF, Lynch M, Mayberg HS, McQuillen PS, Nitkin R, Pascual-Leone A, Reuter-Lorenz P, Schiff N, Sharma A, Shekim L, Stryker M, Sullivan EV, Vinogradov S. Harnessing neuroplasticity for clinical applications. Brain. 2011 Jun;134(Pt 6):1591-609. doi: 10.1093/brain/awr039. Epub 2011 Apr 10. PMID 21482550
- [Background] Sibille KT, Bartsch F, Reddy D, Fillingim RB, Keil A. Increasing Neuroplasticity to Bolster Chronic Pain Treatment: A Role for Intermittent Fasting and Glucose Administration? J Pain. 2016 Mar;17(3):275-81. doi: 10.1016/j.jpain.2015.11.002. Epub 2016 Feb 2. PMID 26848123